# **OBSERVATIONAL STUDY**

Clinical and Economic Outcomes of hs-cTns for diagnosis of NSTEMI in Patients With Chest Pain in EDs in Italy-An Observational Study - TROCAR 2017

No Profit Study: TROCAR 2017

#### **Promoter**

National Institute of Health - Istituto Superiore di Sanità (ISS)
National Centre for Health Technology Assessment - Centro Nazionale per l'Health
Technology Assessment (HTA)
Viale Regina Elena 299
00161 Roma

Version 13\_April\_2017

## **SUMMARY**

This multicenter observational study is a clinical, organizational and economic evaluation of the different quantitative assays of high-sensitivity cardiac troponin in patients with suspected acute myocardial infarction and non-ST-elevation ECG (NSTEMI) at admission at 12 Italian Emergency Departments.

# This document provides a synopsis of the Study Protocol (original in Italian)

## **SYNOPSIS**

| Title | Clinical and Economic Outcomes of hs-cTns for diagnosis of NSTEMI in Patients With Chest Pain in EDs in Italy-An Observational Study TROCAR 2017 |
|---|---|
| Promoter | National Institute of Health National Health Technology Assessment Centre |
| Type of study | No profit with in vitro diagnostic medical devices routinely employed in clinical practice |
| Clinical phase | Post marketing |
| Background | Myocardial infarction is one of the leading causes of death and disability worldwide. In addition to standard diagnostic methods, it has been shown that high-sensitivity cardiac troponin assays allow greater sensitivity in the diagnosis of myocardial infarction and assume a central role for both exclusion ("rule out") and confirmation ("rule in") of acute myocardial infarction, while allowing to reduce the time interval between Emergency Department admission and presumptive diagnosis. |
| | Considering the relevance of this topic, we propose to conduct an observational study in real world clinical practice settings at Emergency Departments, aiming to evaluate clinical and economic aspects deriving from the use of the different quantitative assays of high-sensitivity cardiac troponin currently available in patients with suspected acute myocardial infarction and non-ST-elevation ECG (No ST elevation myocardial infarction - NSTEMI) at admission, including time of diagnosis and number of laboratory and imaging tests performed. |
| Study design | Observational |
| Objective | Clinical, organizational and economic evaluation of the different quantitative assays of high-sensitivity cardiac troponin in patients with suspected acute myocardial infarction and non-ST-elevation ECG (NSTEMI) at admission at the Emergency Department |

| Primary Endpoint | Time to diagnosis at the Emergency Department |
|---|---|
| Secondary Endpoints | % rule in patients (NSTEMI diagnosis) |
| | % rule out patients (exclusion of NSTEMI) |
| | % patients dead 30 days after Emergency Department admission |
| | % patients with myocardial infarction 30 days after Emergency |
| | Department admission |
| | % patients with major adverse events 30 days after ED |
| | admission |
| Pharmacoeconomic | Number and cost of laboratory and imaging tests performed at |
| endpoint | the Emergency Department |
| Evaluation of | Outcome measures: time of diagnosis, death or myocardial |
| effectiveness | infarction 30 days after Emergency Department admission. |
| | Sensitivity and Negative Predictive Value of myocardial Infarction |
| | ("rule out") with different quantitative assays of high-sensitivity |
| | cardiac troponin, according to the standard operating protocols |
| | of the participating Centers. |
| | Sensitivity and Negative Predictive Value will be evaluated in |
| | relation to: |
| | a) limit of detection of the used assay |
| | b) 99th percentile of the reference healthy population |
| | Evaluation of 30-day prognosis |
| | Evaluation of costs of any further examinations after the first |
| Safety evaluation | N.A. (already provided in the Hospital) |
| Expected number of | |
| patients | 300 patients for each centre |
| Type of patients | Patients with suspected acute myocardial infarction and non-ST- |
| l ypo or pationto | elevation ECG (NSTEMI) at admission at the Emergency |
| | Department |
| Type and number of | 12 Emergency Departments |
| centres | |
| Enrollment | Consecutive |
| Number of examinations | Patients will be examined at enrollment in the Emergency |
| | Departments, and after 30-days |
| Inclusion and exclusion | Inclusion criteria |
| criteria | |
| | both sexes |
| | ≥18 years old |
| | Patients with chest pain |
| | At least one high-sensitivity cardiac troponin test |
| | performed |
| | Written informed consent |

| | Exclusion criteria |
|---|---|
| | <ul> <li>Refusal to provide informed consent</li> <li>Elevation of ST segment in the ECG</li> <li>Pregnancy or breastfeeding</li> <li>Any other clinical conditions not compatible with participation at the study</li> </ul> |
| Used in-vitro medical device | Different quantitative assays of high-sensitivity cardiac troponin currently available and used in the Emergency Department |
| Length of study | January 2018 - July 2018 |

#### References

- 1. Thygesen K, Alpert JS, Jaffe AS, Simoons ML, et al. Third Universal Definition of Myocardial Infarction. J Am Coll Cardiol 2012; 60 (16): 1581-1598.
- 2. Roffi M, Patrono C, Collet JP, et al. 2015 ESC Guidelines for the management of acute coronary syndromes in patients presenting without persistent ST-segment elevation. Eur Heart J 2016; 37: 267-315.
- 3. Apple FS, Collinson PO, and for the IFCC Task Force on Clinical Applications of Cardiac Biomarkers. Analytical Characteristics of High-Sensitivity Cardiac Troponin Assays Clin Chem 2012; 58 (1): 54-61.
- 4. Apple FS, Lee R, Murakami MM. Determination of 19 cardiac troponin I and T assay 99th percentile values from a common presumably healthy population. Clin Chem 2012; 58:1574–1581.
- 5. Shah AS, Anand A, Sandoval Y, et al: High-sensitivity cardiac troponin I at presentation in patients with suspected acute coronary syndrome: a cohort study. Lancet 2015; 386: 2481-2488.
- 6. Rubini Gimenez M, Twerenbold R, Jaeger C, et al. One-hour rule-in and rule-out of acute myocardial infarction using high-sensitivity cardiac troponin I. Am J Med 2015; 128: 861-870.
- 7. Shah ASV, Griffiths M, Lee KK, et al. High sensitivity cardiac troponin and the underdiagnosis of myocardial infarction in women: prospective cohort study. BMJ 2015;350:g7873.
- 8. NICE (National Institute for Health and Care Excellence). Myocardial infarction (acute): early rule out using high-sensitivity troponin tests (Elecsys Troponin T high-sensitive, ARCHITECT STAT High Sensitive Troponin-I and AccuTnI+3 assays). NICE diagnostics guidance 15, issued October 2014.
- 9. Casagranda I, Cavazza M, Clerico A, et al. Proposal for the use in emergency departments of cardiac troponins measured with the latest generation methods in patients with suspected acute coronary syndrome without persistent ST-segment elevation. Clin Chem Lab Med 2013; 51: 1727-1737.10. Boeddinghaus J, Reichlin T, Cullen L, et al. Two-

hour algorithm for triage toward rule-out and rule-in of acute myocardial infarction by use of high-sensitivity cardiac troponin I. Clin Chem 2016; 62: 494-504.

- 11. Cremonesi P, Di Bella E, Montefiori M. Cost analysis of emergency department. J Prev Med Hyg 2010; 51: 157-163.
- 12. Keller T, Zeller T, Ojeda F, et al. Serial Changes in Highly Sensitive Troponin I Assay and Early Diagnosis of Myocardial Infarction. JAMA. 2011; 306: 2684-2693.
- 13. Reichlin T, Irfan A, Twerenbold R, et al. Utility of absolute and relative changes in cardiac troponin concentrations in the early diagnosis of acute myocardial infarction. Circulation 2011; 124: 136–145.
- 14. Pickering JW, Greenslade JH, Cullen L, et al. Validation of presentation and 3 h high-sensitivity troponin to rule-in and rule-out acute myocardial infarction. Heart 2016; doi:10.1136/heartjnl-2015-308505.